CLINICAL TRIAL: NCT05417178
Title: Validation of myStrength's Macropersonalization Engine
Acronym: PAG-Macro
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Teladoc Health (Industry)
Responsible Party: Sponsor
Other Study IDs: PAG_Macro 2022
Record Dates: First submitted 2022-05-22; First posted 2022-06-14 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Depression, Anxiety; Trauma
Keywords: Sleep; Digital Therapy
MeSH Terms: conditions — Depression; Anxiety Disorders; Wounds and Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: myStrength Macropersonalization Enginge — An onboarding process that utilizes the PHQ-9, GAD-7, and WHO-5 that leads to a user of the digital program's clinical focus and primary, secondary, and tertiary intervention recommendations.

SUMMARY:
This is a study to validate myStrength's macropersonalization algorithm. Specifically, the study seeks to answer: Does myStrength's macropersonalization algorithm match what a clinician would offer as a diagnosis following an expert assessment? Participants will be treatment-seeking adults, ages 18 to 65, recruited from an evidence-based group psychotherapy practice. Participants will be asked to complete myStrength onboarding and a clinician-conducted initial assessment. Inter-rater reliability will be assessed to determine the consistency between myStrength and clinician in primary focus area of digital program.

DETAILED DESCRIPTION:
Rationale and Background: Macropersonalization refers to the rules applied to a member's onboarding data that dictate their primary clinical focus and available interventions that will be recommended. Macropersonalization is a new myStrength feature that is meant to enable myStrength's ability to deliver evidence-based stepped care.

Research Questions: To examine the inter-rater reliability between myStrength's macropersonalization engine and expert clinical recommendations for members' primary clinical focus.

Study Design: This is a one-arm, prospective study.

Population: Study participants will be adults, ages 18 to 65, seeking therapy at an evidence-based psychotherapy group practice.

Data Sources: Anticipated data sources include members myStrength onboarding data, macropersonalization outputs, and clinician-administered clinical assessments.

Data Analysis: A Cohen's kappa will be generated for agreement between myStrength macro-personalization primary focus area and clinician diagnosis to fulfill the primary objective. Conditional kappas based on stratification, as well as a logistic regression, will be used to determine whether demographics or treatment history are associated with concordance, and qualitative analyes will be used to describe sub-clinical or secondary focus areas associated with clinician diagnoses.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 85, inclusive
* Able to read, write, and speak in English
* Has access to the Internet to complete study procedures
* Currently engaged in therapy or has schedule an initial appointment with the Pacific Anxiety Group

Exclusion Criteria:

* None

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be individuals seeking initial evaluation and treatment at the Pacific Anxiety Group.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Inter-rater reliability on primary focus area | Upon completion of initial assessments by subject and clinician within 30 days of signing informed consent.
  Inter-rater reliability between myStrength macropersonalization engine and expert clinical recommendation for an individual's primary focus

CONTACTS AND LOCATIONS:
Overall Officials: Bobbie James, MStat, Study Director — Teladoc Health
Locations (1):
- Pacific Anxiety Group, Menlo Park, California, United States

IPD SHARING:
Plan to Share IPD: Undecided